CLINICAL TRIAL: NCT02739061
Title: Shanghai Mental Health Center in China
Brief Title: The Study of the Pathogenesis and Cognitive Behavioral Group Therapy in Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYZhang
Record Dates: First submitted 2016-04-12; First posted 2016-04-14 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2018-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: pathogenesis; cognitive behavioral group therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Sertraline; Fluvoxamine; Drug Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- cognitive behavioral group therapy (Active Comparator): cognitive behavioral group therapy
  Interventions: Behavioral: cognitive behavioral group therapy
- drug therapy (Active Comparator): drug therapy
  Interventions: Drug: sertraline, fluvoxamine
- The combination therapy (Active Comparator): cognitive behavioral group therapy and drug therapy
  Interventions: Other: cognitive behavioral group therapy and drug therapy

INTERVENTIONS:
Behavioral: cognitive behavioral group therapy — Establish closed every collection of six or so patients structured group. Each group patients were treated for 12 times, once a week, 120 minutes at a time.
  Treatment for 1 to 3 times to obsessive-compulsive disorder and cognitive behavioral therapy as the theme of psychological education; 4 to 6, 8 to 10 times exposed step by step and reaction treatment and prevention of training;7 and 11 times invite patients family members or other caregivers, make education about obsessive-compulsive disorder cognitive behavioural therapy, to promote patients exposed response prevention homework completion and social support; The 12th time treatment is self assessment and treatment guidelines for a long time.
  Arms: cognitive behavioral group therapy
Drug: sertraline, fluvoxamine — Select specified drugs (sertraline, fluvoxamine)
  Arms: drug therapy
Other: cognitive behavioral group therapy and drug therapy — Select specified drugs (sertraline, fluvoxamine) and start group cognitive behavior therapy for 12 weeks at the same time
  Arms: The combination therapy

SUMMARY:
This study intends to explore the pathogenesis of obsessive-compulsive disorder(OCD) by using biological technologies such as genetics and imaging, and to evaluate the efficacy of group cognitive behavioural therapy in OCD among the Chinese people. We also prepare to explore the synergistic effect of the pharmacological treatment combined with group cognitive behavioural therapy in OCD, and to find the biological and psychological index which can predict curative effect.

This research includes case control study and randomized controlled single-blind study. At baseline, we compare the dimensions of clinical symptoms, genetics and imaging between OCD patients and healthy controls. The OCD patients are randomly assigned into pharmacological treatment, psychological treatment or pharmacological combined with psychological treatment for a 12-week treatment. After a 12-week treatment, the OCD patients will be divided into valid and invalid groups according to the results of our randomized controlled study by researchers: to our valid group, patients will continue the current treatment, and to the invalid psychological or pharmacological treatment group, patients will have a 12-week combined treatment. From the baseline, we will have a 9-month follow up for both OCD patients and healthy controls.

DETAILED DESCRIPTION:
1. Case control study: At baseline, comparing the dimensions of clinical symptoms, genetics and imaging between OCD patients and healthy controls who were chosen into our study.
2. Randomized controlled single-blind study: The OCD patients are randomly assigned into pharmacological treatment, psychological treatment or pharmacological combined with psychological treatment. Psychological treatment: every six or so patients can establish a closed structured group. Each group will be treated for 12 sessions, for once a week, 120 minutes at a time. The 1-3 session will be psychological education on the topic of OCD and cognitive behavioral therapy; The 4-6 and 8-10 session will do step by step exposure and response prevention(ERP) training; the 7th an 11th session will invite family members or other caregivers of OCD patients for a education about OCD cognitive behavioral therapy to facilitate patients to complete ERP homework and give them some social supports; the final session will be self treatment evaluation and long-term treatment guidance. Pharmacological treatment: This study choose the SSRIs(Selective Serotonin Reuptake Inhibitor:sertraline, fluvoxamine, initial dose of 50 mg, the dose can be adjusted once a week, and the maximum dose should under the instruments ) approved by SFDA(China Food and Drug Administration) for OCD treatment which will last 12 weeks. Patients with sleep disorder can combined with Benzodiazepines less than two consecutive weeks; combination with other psychotropic drugs are forbidden. Pharmacological combined with psychological treatment: every six or so patients can establish a closed structured group which is same as the psychological treatment group; patients start to take medicine at the same time, use of the medicine is same as the pharmacological treatment group.
3. Follow-up study: After finishing the 12-week treatment, the OCD patients will be into a 6-month follow-up. Patients who are satisfied with pharmacological and/or psychological treatment will continue the current treatment, while others' follow-up treatment and specific treatment ways will be decided by researchers through the results of of our randomized controlled study. Our randomized controlled study results will be divided into valid and invalid groups. To the invalid psychological or pharmacological treatment group, patients will have a 12-week combined treatment which means invalid pharmacological treatment need to combine with psychological treatment and invalid psychological treatment need to combine with pharmacological treatment. Invalid pharmacological combined with psychological treatment should adjust the medicine (change with sertraline/fluvoxamine) and go on the psychological treatment. After the baseline assessment, OCD patients will have a follow-up evaluation at the 16th, 24th, and 36th week, while the healthy control will have a follow-up evaluation at the 12th and 36th week.

ELIGIBILITY:
Inclusion Criteria:

* OCD patients： Among 18 to 54 years old, males or females； See a doctor because of OCD recently，conform to DSM-Ⅳ(Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria of OCD; The scores of the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) is not less than 16 points; Has not yet accepted psychiatric medication or have received irregular medication treatments and discontinuation for at least eight weeks; A junior high school and above level of education; Has enough of seeing and hearing level to complete the necessary checks; Right-handed (this standard is limited to magnetic resonance imaging (MRI) detection); The Han nationality (this standard is limited to genetic testing); Willing to participate in this study..
* Healthy controls： 1:1 match with the OCD group in age, gender and level of education; Never appear symptoms of OCD, not comply with obsessive compulsive disorder, or other mental disorders DSM-Ⅳ diagnostic criteria; There is no history of psychiatric medication; No two lines three generations of history of mental disorder; Has enough of seeing and hearing level to complete the necessary checks; Right-handed (this standard is limited to magnetic resonance imaging (MRI) detection); The Han nationality (this standard is limited to genetic testing); Willing to participate in this study.

Exclusion Criteria:

* OCD patients： Conform to the DSM-Ⅳ other axis I except obsessive-compulsive disorder diagnosis (M.I.N.I evaluation screening); Patients will not be able to complete the required assessment check and cognitive behavioural therapy because of the severe OCD symptoms; There is negative or a higher risk of suicide; Currently suffering from serious physical disease or central nervous system disease, substance abuse; Pregnant woman or woman who is ready to be pregnant, and lactating women; Used to have received a full course of cognitive behavioral therapy, and no significant curative effect; In presence of metallic implants: install pacemaker, intracranial silver clip, metal false teeth, stents, artery clamp, joints, metal fixed, or other metal implants in (this standard is limited to magnetic resonance imaging (MRI) detection).
* Healthy controls： There is negative or a higher risk of suicide; Currently suffering from serious physical disease or central nervous system disease, substance abuse; Pregnant woman or woman who is ready to be pregnant, and lactating women; In presence of metallic implants: install pacemaker, intracranial silver clip, metal false teeth, stents, artery clamp, joints, metal fixed, or other metal implants in (this standard is limited to magnetic resonance imaging (MRI) detection).

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Y-BOCS (The Yale-Brown Obsessive Compulsive Scale) | up to 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Shen, Senior, Study Director — Shanghai Mental Health Center
Locations (1):
- Clinical psychiatrist, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No